CLINICAL TRIAL: NCT02840747
Title: A Tissue Repository for the Collection of Samples From Patients With Cutaneous T Cell Lymphoma and Healthy Volunteers
Brief Title: Tissue Repository: CTCL Collection Protocol
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAQ8751
Record Dates: First submitted 2016-07-15; First posted 2016-07-21 (Estimated); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Lymphoma, T-Cell, Cutaneous; Lymphomatoid Papulosis; Sézary Syndrome
Keywords: Lymphomatoid Papulosis; Sézary Syndrome; T-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Lymphomatoid Papulosis; Lymphoma, T-Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsies, swabs (skin, cheek epithelium, nasal), samples of blood, fecal and urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with CTCL: Skin biopsies, blood samples, skin swabs, nasal swabs, cheek epithelium swabs, fecal samples and urine samples may be collected from patients with CTCL (according to World Health Organization-European Organization for Research and Treatment of Cancer (WHO-EORTC) criteria).
- Patients with benign dermatoses: Skin biopsies, blood samples, skin swabs, nasal swabs, cheek epithelium swabs, fecal samples and urine samples may be collected from patients with benign dermatoses, including but not limited to conditions such as eczema, psoriasis, and dermatitis.
- Healthy Controls: Skin biopsies, blood samples, skin swabs, nasal swabs, cheek epithelium swabs, fecal samples and urine samples may be collected from healthy volunteers.

SUMMARY:
This document is a protocol for a non-interventional human research study in which the investigator hopes to better understand the changes that take place in T cells in Cutaneous T-cell lymphoma (CTCL). The purpose of this study is to establish a protocol for the collection and storage of tissue samples from patients with CTCL for future research studies. Collection and storage of tissue samples from control patients will also be carried out.

DETAILED DESCRIPTION:
CTCL is a heterogeneous group of non-Hodgkin's lymphomas characterized by chronic inflammation and accumulation of malignant T cells in the skin. In order to carry out research to expand the knowledge and develop more effective treatments, tissue samples from CTCL patients with presumed or known disorders are required and tissue samples from control patients will be required to compare the differences between affected and healthy populations.

Scientists will be able to test new ideas and new technologies that are not apparent or available at the present moment from this tissue repository in the future. This type of information will thus be of great advantage to future patients with these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CTCL or Lymphomatoid Papulosis (LYP): a clinical or histologic diagnosis of a) newly diagnosed, b) progressive, or c) relapsed CTCL or LYP who are initiating or changing therapy.
* Patients with Sézary Syndrome (SS) or stage IV B CTCL as defined by blood involvement on flow cytometry or morphology: (1) ≥1000/μL Sézary cells by morphology; (2) Cluster of differentiation 4 (CD4)/cluster of differentiation 8 (CD8) ratio ≥10; (3) CD4+cluster of differentiation 7 (CD7)- cells ≥40 percent; (4) or CD4+cluster of differentiation 26 (CD26)- cells ≥30 percent.
* Ability to understand and willing to sign a willing informed consent document.
* Age ≥ 18 years.

Inclusion Criteria for Age and Sex Matched Controls:

* Matched for sex, and age +/- 10 years.
* Ability to sign informed consent document.
* Patients with or without benign inflammatory skin conditions including, but not limited to, eczema, psoriasis, or dermatitis or Patients without skin conditions requiring treatment with systemic immunosuppressive, biologic, or chemotherapeutic agents.

Exclusion Criteria:

* Patients with a history of previous lymphoma other than CTCL or SS or LYP.
* Medical illnesses with potential suppressive or activating impact on immune and bowel function as judged by the investigator.
* Current, viable pregnancy.
* Anemia with a documented hemoglobin laboratory value of <7.5 g/dl within the past 6 months.

Exclusion Criteria for Age and Sex Matched Controls:

* Previous history of CTCL, SS, LYP, or any lymphoma.
* Previous history of Human Immunodeficiency Virus (HIV) infection.
* Anemia with a documented hemoglobin laboratory value of <7.5 g/dl within the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This protocol is for the collection of biological specimens from patients who fall into the following three groups:
  1. Patients with diagnosis of cutaneous T cell lymphoma (diagnosed according to the WHO-EORTC criteria)
  2. Patients with benign dermatoses, including but not limited to psoriasis, eczema, and dermatitis.
  3. Healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-07; Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of biological specimen collections | 2 years
  This is a collection protocol to establish a tissue repository for samples from patients with CTCL.

CONTACTS AND LOCATIONS:
Overall Officials: Larisa J. Geskin, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided